CLINICAL TRIAL: NCT01464203
Title: Randomized Controlled Trial to Evaluate the Cost and Clinical Effectiveness of CT Coronary Angiography in Patients With Stable Angina Pectoris (RADICAL Trial)
Brief Title: Role of Cardiac CT in Rapid Access Chest Pain Clinics (RADICAL)
Acronym: RADICAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: AJAY YERRAMASU (Other Government)
Collaborators: Wellington Hospital (Other Government); Barnet and Chase Farm Hospitals NHS Trust (Other); Chase Farm Hospital (Other); Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor-Investigator, AJAY YERRAMASU, Clinical Research Fellow, Wellington Hospital
Organization: Wellington Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RADICAL Trial
Record Dates: First submitted 2011-10-15; First posted 2011-11-03 (Estimated); Last update posted 2011-11-03 (Estimated); Status verified 2011-10

CONDITIONS: Coronary Artery Disease
Keywords: Computed tomographic coronary angiography; multi-slice CT; angina; cost-effectiveness
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CT coronary angiography (Experimental): Patients in this arm will undergo CT coronary angiography to assess the patency of coronary arteries and their clinical management will be decided by the results of CT coronary angiography.
  Interventions: Other: CT coronary angiography
- Control Arm (Active Comparator): Patients in this arm will receive the "standard of care" (SoC). They will undergo either coronary angiography, myocardial perfusion scan or stress echocardiography as decided by the physician in charge, depending on the local availability of individual investigations and the patient's clinical scenario.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: CT coronary angiography — CT coronary angiography:
  This allows two distinct assessments of the coronary arteries to be made:
  * coronary calcium scan, which is a 30 second, low-radiation scan that allows reproducible quantification of the amount of calcium in the coronary arteries to be made.
  * contrast enhanced CT coronary angiogram. This is a quick, non-invasive scan to assess the patency of coronary arteries.
  Arms: CT coronary angiography
Other: Standard of Care — The management of patients in this group is according to the NHS protocol and is not altered by their participation in the trial. The choice of diagnostic investigation for CAD is determined by the patient's clinical scenario and the availability of different diagnostic modalities in the recruiting hospital.
  Arms: Control Arm

SUMMARY:
Heart disease remains the most common cause of death in the UK. Chest pain is often the first presenting symptom in patients with heart disease, and may be a warning signal prior to a heart attack or death. The diagnosis based on symptoms alone however is unreliable and further testing is almost always necessary.

Rapid access chest pain clinics (RACPCs) are able to expedite the assessment of such patients. The principal investigation used is an exercise stress electrocardiogram (s-ECG). Although simple, cheap, and convenient, the s-ECG is often inaccurate; missing the diagnosis or falsely suggesting the diagnosis. This can happen in as many as 25% of patients, resulting in a delay in treatment or unnecessary further investigation.

CT Angiography (CTA) is a novel non-invasive technique where the coronary arteries can be visualised by Computerised Tomography. In previous studies it shows a high degree of correlation with invasive angiography, with a high accuracy for the diagnosis of obstructive coronary artery disease. However, the technique is relatively new, and its full role is yet to be defined in the clinical setting of a chest pain clinic. The investigators do not at present have any information as to whether it is able to speed up the diagnosis, reduce the need for other tests, and therefore also costs.

In this trial, the investigators aim to examine the accuracy and cost effectiveness of CTA in patients with suspected cardiac chest pain presenting to a chest pain clinic, when compared to the more established techniques like s-ECG, myocardial perfusion scanning and coronary angiography. The study will enable us to establish the optimal and most cost effective strategy for investigation of patients presenting to chest pain clinics.

DETAILED DESCRIPTION:
Study Objectives:

* To assess the diagnostic accuracy and cost effectiveness of non-invasive coronary angiogram by Cardiac CT in the diagnosis of coronary artery disease in patients with angina, in the setting of Rapid Access Chest Pain clinics
* To formulate an optimal diagnostic algorithm in terms of accuracy and cost effectiveness for diagnosis of CAD in patients with chest pain.

Study Setting:

- Rapid Access Chest Pain clinics in 3 NHS hospitals (Barnet, Chase Farm and the Royal Free hospitals)

Target Population:

- Patients with new onset, stable exertional angina presenting to Rapid Access Chest Pain clinics.

Study Design and Methodology:

This trial is designed as a prospective randomized case - control study. 600 patients who meet the study criteria will be recruited from Rapid Access Chest Pain Clinics. The patients will be randomized into 2 cohorts (study and control) of 300 each. All patients will undergo stress - ECG at the referring hospital. Patients in the control group will receive the 'standard clinical care'. Their management is not altered by their inclusion in the trial. All patients in the study group will undergo CT coronary Angiography at the Clinical Imaging and Research Centre based at the Wellington Hospital. Patients with obstructive coronary artery disease (defined as >50% stenosis in left main coronary artery or >70% stenosis in one of the other major epicardial coronary arteries) will be referred for invasive coronary angiography +/- revascularization. Patients with intermediate (50-70%) coronary stenosis will be referred to myocardial perfusion scan (MPS). Patients with significant reversible ischemia on MPS will be referred to invasive coronary angiography +/- revascularization. Patients who do not have evidence of significant reversible ischemia on MPS and those with <50% stenosis on CT coronary angiogram will be discharged on appropriate medications. All patients will be followed up for 12 months after recruitment. Information will be gathered regarding clinical events (non-fatal/fatal MI, acute coronary syndrome, hospitalization, emergency/elective revascularization) and quality of life as per SF-36 questionnaire. All the diagnostic and therapeutic procedures underwent by each patient in both cohorts will be recorded. The cost-effectiveness of each CT coronary angiography will be calculated by using the NHS reference costs.

Primary outcome measure: The total cost of diagnosis for current diagnostic strategy being used in the Rapid Access Chest Pain Clinics and a new strategy involving the use of CT coronary angiography in the investigation of patients with angina.

Secondary outcome measures:

* Diagnostic Accuracy of CT coronary angiography
* Prognostic value of CT coronary angiography
* Number of normal angiograms in each cohort
* Number of angiograms not followed by revascularization in each cohort
* Quality of life as assessed by SF-36 Questionnaire

For calculating cost effectiveness, NHS reference costs will be used. Thus, the costs and benefits will be considered from the NHS perspective

ELIGIBILITY:
Inclusion Criteria:

* chest pain or shortness of breath suspected to be due to coronary artery disease

Exclusion Criteria:

* Age < 40 years
* Pregnancy
* Serum Creatinine > 150 mmol/L or eGFR < 40
* Established or suspected acute coronary syndrome
* Previous history of PTCA
* Atrial Fibrillation
* History of allergy to iodinated contrast media

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Cost of diagnosis | one year

SECONDARY OUTCOMES:
Diagnostic Accuracy of CT coronary angiography | one year
  Diagnostic accuracy of CT coronary angiography in detecting >50% coronary stenosis, using invasive coronary angiography as reference standard.
Quality of life | one year
  quality of life is measured in the study and control subjects after a median follow-up period of one year, using SF-36 questionnaire
Number of normal invasive coronary angiograms | one year
  Number of invasive coronary angiograms that show either normal coronary arteries or non-obstructive coronary disease (<50% coronary stenosis) will be measured and compared between study and control groups
Number of invasive coronary angiograms not followed by coronary revascularization | one year
  Number of invasive coronary angiograms that are not followed by revascularization will measured and compared between study and control groups.
Prognostic value of CT coronary angiography | 1 year
  Prognostic value of CT coronary angiography in predicting major adverse cardiovascular events over a median follow-up period of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Deven Patel, MBBch, FRCP, Principal Investigator — Barnet Hospital, Wellhouse Lane, Barnet, UK
Locations (3):
- United Kingdom (3):
  - Barnet and Chase Farm Hospitals NHS Trust, Barnet, Hertfordshire
  - Royal Free Hospital NHS Trust, London, London
  - Clinical Imaging and Research Centre, Wellington Hospital, London, London

REFERENCES:
- [Background] Yerramasu A, Venuraju S, Lahiri A. Evolving role of cardiac CT in the diagnosis of coronary artery disease. Postgrad Med J. 2011 Mar;87(1025):180-8. doi: 10.1136/pgmj.2009.093815. Epub 2010 Aug 5. PMID 20693150
- [Derived] Yerramasu A, Lahiri A, Venuraju S, Dumo A, Lipkin D, Underwood SR, Rakhit RD, Patel DJ. Diagnostic role of coronary calcium scoring in the rapid access chest pain clinic: prospective evaluation of NICE guidance. Eur Heart J Cardiovasc Imaging. 2014 Aug;15(8):886-92. doi: 10.1093/ehjci/jeu011. Epub 2014 Feb 9. PMID 24513880